CLINICAL TRIAL: NCT06600685
Title: Functionally Oriented Music Therapy (FMT) In The Treatment Of Long Term Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mälardalen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-04082-01
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Long Term Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Phase 1.) Single case research experimental design. N=10 participants will be asked to answer a set of questionnaires (Lickert-scales) every week for three weeks before the start of the treatment period and after completing FMT sessions 2, 4, 6, 8, and 10. This is to capture results based on patients' self-assessments during entire FMT treatment. Three measurement sessions will be completed before treatment begins to capture the baseline of their condition and pain in their daily life. Participants will begin their measurements on different weeks, to reduce the risk that the baseline measurement is due to any external factors that may affect participants if they are measured during the same time period/week.
  Phase 2.) Pilot study with a mixed design. Relevant outcome measures (from phase 1) will be used to achieve valid and reliable results. N=60 participants will be recruited to participate in FMT treatment during a period of ten weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT arm (Other)
  Interventions: Other: Functionally oriented music therapy (FMT)

INTERVENTIONS:
Other: Functionally oriented music therapy (FMT) — There are different methods of music therapy and one of these is FMT. It is a body-based and music therapeutic treatment method that is used for health-promoting purposes. With the help of i.e. drums, cymbals, various custom-made drumsticks, flutes, chairs, balance balls and balance cushions. FMT strives to support, strengthen and develop the person's physical, mental and social abilities. FMT-sessions (20 minuets/1 time a week) are performed individuelly (a patient with a educated music therapist).

SUMMARY:
Project idea: This project aims to explore and evaluate a hitherto unexplored treatment method for people living with long-term musculoskeletal pain. The project's starting point is that it is urgent to develop evidence-based methods that can promote health and well-being, alleviate suffering and lead to an improved quality of life in the target group. The method "Functionally oriented music therapy" (FMT), to be studied in the present project, can be such a method. In FMT, music and movement are combined for health-promoting purposes, which can be assumed to lead to experiences of well- being and recovery. The method is already used in primary care in Region Sörmland, but the method is not evidence-based in the treatment of long-term musculoskeletal pain, which is why scientific evaluation is needed. The project is urgent both from a societal and patient perspective, among other things because healthcare resources need to be used more efficiently than today. To evaluate the method, both qualitative and quantitative research methodology will be used. If the results of the project are positive, i.e., if we can find evidence that various aspects of health are specifically affected/improved, then the results can contribute to evidence based FMT support for health promotion purposes for people with long-term musculoskeletal pain. If, on the other hand, the results show that FMT has no or only little effect, that in itself is an important contribution to new knowledge about treatment and recovery in people with long-term musculoskeletal pain. Today, FMT is used in, among other things, habilitation, rehabilitation and psychiatric care. However, research is needed that deals with the method's health-promoting efforts even in the case of long-term musculoskeletal pain problems.

ELIGIBILITY:
Inclusion Criteria:

* People with long-term musculoskeletal pain that occurred for at least three months.
* People over 18 years of age.
* People able to understand and speak Swedish or English

Exclusion Criteria:

* Severe hearing loss
* Visual impairment
* Cognitive impairment.

Pain conditions caused by:

* malignancy
* severe spinal pathology or
* neurological disease that severely limit the ability to perform activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Improved quality of life | Assessed every 2 weeks for 10 weeks.
  Support, strengthen and develop the person's physical, mental and social abilities. Questionnaires concerning; body awareness, pain level, management of pain and fear of movement, pain-related activity limitations, emotions, depressive symptoms and anxiety, self-reported sick-leave and general perceived health will be used. The questionnaires are validated and psychometrically evaluated. Self-estimation (using different Lickert-scales).
  The results of phase 1 can contribute to the addition of more outcome measures in phase 2.

CONTACTS AND LOCATIONS:
Locations (1):
- FMT centrum, Eskilstuna, Eskilstuna, Sweden

IPD SHARING:
Plan to Share IPD: No